CLINICAL TRIAL: NCT05625529
Title: Exoluminate Study: Observational Registry Study to Assess Exo-PDAC Assay Performance for Detection of Pancreatic Adenocarcinoma (PDAC) in High-Risk or Clinically Suspicious Patients
Brief Title: ExoLuminate Study for Early Detection of Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: Biological Dynamics (Industry)
Responsible Party: Principal Investigator, Harmeet Dhani, Medical Director, Biological Dynamics
Other Study IDs: BioDyn-011
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Pancreas Cancer; Exosomes; Extracellular Vesicles; Pancreatic Neoplasms
Keywords: Early Detection; Exosomes; Extracellular Vesicles; IPMN; PDAC; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Double-spun plasma, EDTA tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- Cohort 1: Individuals without history of PDAC meeting any of the following criteria:
  A. 2+ relatives with PDAC on same side of family; 2 are first degree related to each other and at least 1 is first degree related to subject; age ≥ 50 years or ≤10 years younger than earliest PDAC in family at diagnosis.
  B. 2+ first degree relatives with PDAC; age ≥ 50 years or ≤ 10 years younger than earliest PDAC in family at diagnosis.
  C. BRCA1, BRCA2, PALB2, ATM, MLH1, MSH2, MSH6, PMS2, EPCAM pathogenic or likely pathogenic variant AND 1 first or second degree relative with PDAC; age ≥ 50 years or ≤ 10 years younger than earliest PDAC in family at diagnosis.
  D. Familial Atypical Moles and Malignant Melanoma (FAMMM) with pathogenic or likely pathogenic CDKN2A variant; age ≥ 40 years.
  E. Peutz-Jegher syndrome with STK11 pathogenic or likely pathogenic variant; age ≥35 years.
  F. Hereditary pancreatitis with PRSS1 pathogenic or likely pathogenic variant and history of pancreatitis; age ≥ 40 years.
- Cohort 2: Individuals without history of PDAC meeting any of the following criteria:
  A. ATM, BRCA1, BRCA2, or PALB2 pathogenic or likely pathogenic variant regardless of family history; age ≥50 years.
  B. Two or more (2+) relatives with PDAC on the same side of family, any degree of relation, not meeting other criteria above; age ≥50 years or ≤10 years younger than earliest PDAC in family at time of diagnosis.
  C. One (1) first degree relative with PDAC at age ≤45 years; ≤10 years younger than PDAC diagnosis in family member at time of diagnosis.
- Cohort 3: A. Individuals meeting criteria for Cohorts 1 or 2 EXCEPT age (i.e. too young to qualify for Cohorts 1 or 2); age ≥ 18 years.
- Cohort 4: A. Individuals without history of PDAC presenting for evaluation who do not meet any criteria for the other cohorts after collection of full family history and/or germline testing, eg. they have only 1 relative with PDAC; age ≥ 18 years.
- Cohort 5 - Personal history of PDAC: Individuals with a personal history of PDAC meeting any of the following criteria (age ≥ 18 years for all subgroups):
  A. Family history includes at least one first degree relative with PDAC, or 2 relatives with PDAC who are first degree related to each other.
  B. Personal or family history of a pathogenic or likely pathogenic germline variant in ATM, BRCA1, BRCA2, CDKN2A, EPCAM, MLH1, MSH2, MSH6, PALB2, PMS2, PRSS1, STK11.
  C. Diagnosed with PDAC at ≤ age 45.
- Cohort 6 - Pancreatic cysts: Individuals with pancreatic cysts (age ≥ 18 years for all subgroups):
  A. Individuals with a pancreatic cystic neoplasm (IPMN) and/or mucinous cystic neoplasm (MCN) and/or PanIN not meeting any criteria for Cohorts 1-3 or 6 (no personal history of PDAC, no known family history of PDAC, no known pathogenic germline variants linked to PDAC risk present in cohorts 1C, 2A, 1D, 1E, and 1F).
  B. Individuals with a pancreatic cystic neoplasm (IPMN) and/or MCN and/or PanIN without PDAC and with at least one of the pathogenic or likely pathogenic gene mutations present in cohorts 1C, 2A, 1D, 1E, and 1F and/or a first degree relative with PDAC.
- Cohort 7 - Acute or chronic pancreatitis: Individuals with a personal history of pancreatitis meeting any of the following criteria (age ≥ 18 years for all subgroups):
  A. Chronic pancreatitis. B. At least 2 episodes of acute pancreatitis.
- Cohort 8 - PDAC stages I-II or clinical suspicion: Individuals with one of the following conditions and treatment naïve (age ≥ 18 years for all subgroups):
  A. Biopsy-proven, clinical stage I-II PDAC and candidate for surgical resection.
  B. Clinical findings suspicious for early stage PDAC prior to biopsy.

SUMMARY:
ExoLuminate is a nationally-enrolling registry study designed for earlier detection of cancer in patients at elevated risk or clinically-suspicious for pancreatic ductal adenocarcinoma (PDAC).

Those with elevated risk for PDAC can include individuals with intraductal papillary mucinous neoplasms, family history of pancreatic cancer, germline mutations in genes known to be associated with cancer, and a personal or family history of pancreatitis.

The goal of the study is to compare the performance of ExoVerita™ assay in early detection of PDAC to current standard-of-care methods of surveillance.

DETAILED DESCRIPTION:
Biological Dynamics, Inc. has developed a non-invasive blood test ("liquid biopsy") that can identify early-stage disease with high sensitivity and specificity. The proprietary ExoVerita™ assay uses alternating current electric (ACE) field to isolate extracellular vesicles (EVs) for differentiated multiomics applications and includes an optimized machine learning algorithm to identify a panel of EV-bound protein biomarkers in patient's plasma in order to detect PDAC at earlier stages.

ExoLuminate is a prospective, multi-center, observational registry study designed to evaluate the non-inferiority of the performance of the ExoVerita™ assay in detecting pancreatic ductal adenocarcinoma (PDAC) in high-risk or clinically-suspicious populations in comparison to standard-of-care methods.

The study is planned to recruit a minimum of 1000 U.S. adults over 3-years (with a 2-year follow-up for data collection).

Eligible subjects will be evaluated using the ExoVerita™ assay through blood donation(s) at specified time intervals. Overall, this study poses minimal risk to subject.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* Meeting criteria for one of the study cohorts.
* Capable of giving informed consent.
* Able to provide a blood sample.

Exclusion Criteria:

* < 18 years old.
* Pregnancy.
* Active cancer (other than pancreatic cancer) and/or undergoing treatment for an active cancer diagnosis (except for skin malignancies).
* Prior organ transplant or bone marrow transplant.
* History of fainting or other adverse effects when blood is drawn.
* Any condition that, in the opinion of the investigator, should preclude enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals at high risk of pancreatic cancer or with stage I-II pancreatic cancer (or clinical suspicion). See cohorts under Groups and Interventions for details.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of ExoVerita™ assay | 36 months or until diagnostic resolution
  Specificity

SECONDARY OUTCOMES:
Clinical performance of ExoVerita™ assay | 36 months or until diagnostic resolution
  Sensitivity
Stage Shift | 36 months or until diagnostic resolution
  Evaluation of stage distribution (SEER) at diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Harmeet Dhani, MD, M.Sc, Principal Investigator — Biological Dynamics
Locations (1):
- Biological Dynamics, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hinestrosa JP, Kurzrock R, Lewis JM, Schork NJ, Schroeder G, Kamat AM, Lowy AM, Eskander RN, Perrera O, Searson D, Rastegar K, Hughes JR, Ortiz V, Clark I, Balcer HI, Arakelyan L, Turner R, Billings PR, Adler MJ, Lippman SM, Krishnan R. Early-stage multi-cancer detection using an extracellular vesicle protein-based blood test. Commun Med (Lond). 2022 Mar 17;2:29. doi: 10.1038/s43856-022-00088-6. eCollection 2022. PMID 35603292
- [Background] Hinestrosa JP, Sears RC, Dhani H, Lewis JM, Schroeder G, Balcer HI, Keith D, Sheppard BC, Kurzrock R, Billings PR. Development of a blood-based extracellular vesicle classifier for detection of early-stage pancreatic ductal adenocarcinoma. Commun Med (Lond). 2023 Oct 19;3(1):146. doi: 10.1038/s43856-023-00351-4. PMID 37857666